CLINICAL TRIAL: NCT00265499
Title: Skeletonized Versus Non-Skeletonized Internal Thoracic Artery Harvest for Coronary Artery Bypass Grafting
Brief Title: The Internal Thoracic Artery Skeletonization Study: A Paired, Within-Patient Comparison
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: R03-41
Record Dates: First submitted 2005-12-13; First posted 2005-12-14 (Estimated); Last update posted 2005-12-14 (Estimated); Status verified 2005-11

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Bypass; Skeletonization; Internal Thoracic Artery; Flow; Length; Pain
MeSH Terms: conditions — Coronary Artery Disease; Pain

INTERVENTIONS:
Procedure: Skeletonization of the internal thoracic artery

SUMMARY:
The purpose of this study is to determine whether skeletonization of the internal thoracic artery leads to improved flow, increased length, improved sternal perfusion, and decreased pain and dysesthesia in patients undergoing coronary artery bypass surgery

DETAILED DESCRIPTION:
Traditional harvesting of the internal thoracic artery (ITA) for use as a conduit in coronary bypass surgery involves the dissection of a rim of tissue surrounding the artery on either side. Although the benefits of ITA use are well established, there are certain limitations to its routine use. Recent studies, primarily observational, have suggested that skeletonization of the ITA (i.e. harvesting of the ITA alone) may overcome some of these limitations by improving conduit flow, increasing length, and reducing the risk of deep sternal infection in high risk patients. Furthermore, skeletonization of the ITA can potentially preserve intercostal nerves and reduce post-operative pain and dysesthesias associated with ITA harvesting. In order to assess the effects of ITA skeletonization, this is a prospective, randomized, within-patient study design in patients undergoing coronary artery bypass grafting.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing bilateral internal thoracic artery harvest for coronary artery bypass surgery

Exclusion Criteria:

* Inability to speak English or French
* Inability to complete follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48

PRIMARY OUTCOMES:
Intra-operative Internal Thoracic Artery Flow measure prior to coronary anastomoses

SECONDARY OUTCOMES:
- Internal Thoracic Artery length
- Sternal Perfusion (SPECT imaging)
- Post-operative pain and dysesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Fraser D. Rubens, MD, Principal Investigator — University of Ottawa Heart Institute, Division of Cardiac Surgery
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada